CLINICAL TRIAL: NCT03235245
Title: Combination of Targeted Therapy (Encorafenib and Binimetinib) Followed by Combination of Immunotherapy (Ipilimumab and Nivolumab) vs Immediate Combination of Immunotherapy in Patients With Unresectable or Metastatic Melanoma With BRAF V600 Mutation : an EORTC Randomized Phase II Study (EBIN)
Brief Title: Immunotherapy With Ipilimumab and Nivolumab Preceded or Not by a Targeted Therapy With Encorafenib and Binimetinib
Acronym: EBIN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1612-MG; 2017-002887-42 (EudraCT Number)
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Unresectable Stage III Melanoma; Stage IV Melanoma
Keywords: cutaneous melanoma; mucosal melanoma; BRAF mutation
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab; encorafenib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: Nivolumab + Ipilimumab (Active Comparator): nivolumab 3 mg/kg q3w + ipilimumab 1 mg/kg q3w for 4 injections followed by nivolumab 480 mg IV q4w until completion of 2 years total treatment or progression. Then treatment will be left at the investigator choice and continued until the 2nd progression.
  Interventions: Drug: Nivolumab + Ipilimumab
- ARM B: Encorafenib + Binimetinib + Nivolumab + Ipilimumab (Experimental): encorafenib 450 mg QD + binimetinib 45 mg BID orally for 12 weeks followed, after a week of pause, by nivolumab 3 mg/kg q3w + ipilimumab 1 mg/kg q3w for 4 injections, followed by nivolumab 480 mg IV q4w until completion of 2 years total treatment or progression. Then patients will be rechallenged with encorafenib 450 mg QD + binimetinib 45 mg BID orally continuously until the 2nd progression.
  Interventions: Drug: Nivolumab + Ipilimumab; Drug: Encorafenib + Binimetinib

INTERVENTIONS:
Drug: Nivolumab + Ipilimumab — nivolumab 3 mg/kg q3w + ipilimumab 1 mg/kg q3w for 4 injections followed by nivolumab 480 mg IV q4w until completion of 2 years total treatment or progression.
Drug: Encorafenib + Binimetinib — encorafenib 450 mg QD + binimetinib 45 mg BID orally for 12 weeks
  Arms: ARM B: Encorafenib + Binimetinib + Nivolumab + Ipilimumab

SUMMARY:
This is a multicenter, 2-arm open-label, randomized comparative phase II study. The objective of this trial is to prospectively evaluate whether a sequential approach with an induction period of 12 weeks with encorafenib + binimetinib followed by combination immunotherapy with nivolumab + ipilimumab improves progression free survival compared to combination immunotherapy nivolumab + ipilimumab alone in patients with BRAF V600 mutation-positive unresectable or metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable stage III or IV cutaneous or mucosal melanoma
* Presence of BRAF V600E or V600K mutation in tumor tissue prior to enrolment as per local assessment
* Tumor tissue from an unresectable or metastatic site of disease must be provided for biomarker analyses. This can be an archived sample if obtained at maximum 3 months prior to randomization and if the patient did not receive treatment since then.
* Measurable disease per RECIST 1.1 criteria by computed tomography (CT) or Magnetic Resonance Imaging (MRI) of Chest/Abdomen/Pelvis CT and brain CT/MRI performed within 28 days prior to randomization
* Patients ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Patients must be able to swallow and retain oral tablets
* Adequate organ function within 14 days prior to randomization
* Patients with hyperthyroidism or hypothyroidism but that are stable on hormone replacement can be included.
* Adequate cardiac function

Exclusion Criteria:

* Uveal melanoma
* Any symptomatic brain or leptomeningeal disease. Subjects with brain metastases are eligible if these have been locally treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment and treatment is completed within 28 days prior to first dose of study drug administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* Any prior treatment for advanced disease including treatment with an anti-Programmed Death receptor-1 (PD-1), anti-Programmed Death-1 ligand-1 (PD-L1), anti-PD-L2, anti-cytotoxic T lymphocyte associated antigen-4 (anti-CTLA-4) antibody, anti-LAG-3, anti-TIM-3, anti-IDO, etc or BRAF or MEK inhibitors.
* History of hypersensitivity to study drugs or any excipient (refer to Investigator's brochures for binimetinib and encorafenib and SmPCs for ipilimumab and nivolumab).
* Prior adjuvant melanoma therapy with IFN, anti-PD1, anti-PDL1 or anti-CTLA-4 or any other systemic treatment is permitted if completed at least 1 year prior to randomization and all related adverse events have either returned to ≤ 1.
* Concomitant administration of strong inducers and inhibitors of P-gp, glucuronidation, CYP3A4 (e.g. rifampicin, rifabutin, carbamazepine, phenytoin or St John's Wort [hypericin])
* Concomitant anticoagulation at therapeutic doses with oral anticoagulants (eg, warfarin)
* Live vaccines within 30 days prior to the first dose of study therapy. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, H1N1 flu, rabies, BCG, and typhoid vaccine.
* Current participation or treatment with other investigational agent or use of an investigational device within 4 weeks of the first dose of study treatment
* Child-Pugh B/C and patients with history of acute or chronic pancreatitis
* Known history or current evidence of active Hepatitis B (e.g., HBsAg reactive) or C (e.g., HCV RNA [qualitative] is detected) or Human Immunodeficiency Virus (HIV) (HIV-1/2 antibodies)
* Chronic use of immunosuppressive agents and/or systemic corticosteroids or any use in the last 15 days prior to the first dose of study treatment
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Autoimmune paraneoplastic syndrome requiring immunosuppressive or dedicated treatment. A specific attention should be given in order to detect any minor myasthenia signs at enrolment; acetylcholine receptor antibodies will be systematically tested when symptoms are suggestive of a myasthenia
* History of any other hematologic or primary solid tumor malignancy, unless in remission for at least 5 years. A patient with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ or pT1a incidental prostate cancer is eligible
* Previous allogeneic tissue/solid organ transplant
* Active infection requiring therapy
* Major surgery or trauma within 12 weeks prior to first dose of treatment or presence of any non-healing wound. Complete wound healing from major surgery must have occurred one month before the first dose of study treatment.

Minor surgery (including uncomplicated tooth extractions) within 28 days before randomization with complete wound healing at least 10 days before randomization is permitted.

* Any anticancer treatment within 4 weeks before randomization e.g. radiation, surgery, systemic therapy.
* Patients with clinically relevant ongoing complications from prior anticancer therapies.
* Severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study, or which would jeopardize compliance with the protocol
* History or current evidence of retinal vein occlusion (RVO) or current risk factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); an ophthalmological assessment is mandatory within 28 days from the first dose of study treatment.
* History of retinal degenerative disease
* Impaired gastrointestinal function or disease that may significantly alter the absorption of encorafenib or binimetinib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption)
* Patients with neuromuscular disorders that are associated with CK > ULN (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. Note: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on binimetinib treatment
* Impaired cardiovascular function or clinically significant cardiovascular diseases
* Uncontrolled hypertension defined as persistent elevation of systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100mmHg, despite current therapy
* History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤ 12 months prior to starting study treatment
* History of thromboembolic or cerebrovascular events ≤ 6 months prior to starting study treatment, including stroke, transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis, pulmonary emboli, aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 4.1 years from first patient in
  PRS is defined as the time from the date of randomization until the first date of progression, or until date of death (whatever the cause), whichever occurs first. Progression will be assessed according to the RECIST criteria (version 1.1)

SECONDARY OUTCOMES:
Overall Survival (OS) | 6 years from first patient in
  OS is defined as the time from the date of randomization to the date of death, whatever the cause.
Complete Response (CR) rate | 4.1 years from first patient in
  CR will be assessed according to the RECIST criteria (version 1.1)
Time to Complete Response (CR) | 4.1 years from first patient in
  Time to CR is defined as the time from the date of randomization until the occurrence of first CR.
Duration of Complete Response (CR) | 4.1 years from first patient in
  Duration of CR will be measured from the time measurement criteria for CR are first met until the first date that recurrence is objectively documented.
Best overall response rate | 4.1 years from first patient in
  Best overall response will be assessed according to the RECIST criteria (version 1.1)
Time to best response | 4.1 years from first patient in
  Time to best response is defined as the time from the date of randomization until the occurrence of the best response (CR or PR, whichever comes first). CR and PR will be assessed according to the RECIST criteria (version 1.1)
Duration of best response | 4.1 years from first patient in
  Best response duration will be measured from the time measurement criteria for CR/PR (whichever is first recorded) are first met until the first date that recurrent or progressive disease is objectively documented. CR and PR will be assessed according to the RECIST criteria (version 1.1)
Occurrence of adverse events | 4.1 years from first patient in
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, for adverse event reporting.
Progression-free survival 2 (PFS2) | 4.1 years from first patient in
  PFS2 is defined as the time from randomization to second objective disease progression, or death from any cause, whichever first. The second objective disease progression will be assessed according to the RECIST criteria (version 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Robert, Principal Investigator — Cancer Institute Gustave Roussy
Locations (38):
- Denmark (2):
  - University Hospitals Copenhagen - Herlev Hospital - University Copenhagen, Herlev
  - Odense University Hospital, Odense
- Finland (2):
  - Helsinki University Central Hospital - Dept of Oncology, Helsinki
  - Tampere University Hospital, Tampere
- France (17):
  - CHU Amiens - Hopital Sud, Amiens
  - CHRU de Besançon - Hopital Jean Minjoz, Besançon
  - CHU de Bordeaux - Groupe Hospitalier Saint-André - Hopital Saint-Andre, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU de Dijon - Centre Georges-François-Leclerc, Dijon
  - CHU de Grenoble - La Tronche - Hôpital A. Michallon, Grenoble
  - CHRU de Lille, Lille
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Leon Berard, Lyon
  - Assistance Publique - Hopitaux de Marseille - Hôpital de La Timone (APHM), Marseille
  - CHU de Nice - Hopital De L'Archet, Nice
  - Assitance Publique - Hopitaux de Paris - Hopital Saint-Louis, Paris
  - CHU Ambroise Pare, Paris
  - Centre Hospitalier De Pau, Pau
  - CHU de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - CHU de Tours - Hopital Trousseau, Tours
  - Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Univ. Mainz - Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz-University Medical Center, Mainz
  - Universitaetsklinikum Wuerzburg, Würzburg
- Italy (7):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - IRCCS - Istituto Oncologico Veneto, Padua
  - IRCCS-Regina Elena National Cancer Center, Roma
  - Universita Degli Studi Di Siena -Policlinico "le Scotte", Siena
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Turin
  - Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia" di Udine, Udine
- The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam, Netherlands
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- Spain (3):
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Badalona
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Vall d'Hebron Institut d'Oncologia, Barcelona
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - East & North Hertfordshire NHS Trust - East and North Hertfordshire NHS Trust - Mount Vernon Hospital, Middlesex

IPD SHARING:
Plan to Share IPD: Yes
All publications must comply with the terms specified in the EORTC Policy 009 "Release of Results and Publication Policy".

REFERENCES:
- [Derived] Robert C, Kicinski M, Dutriaux C, Routier E, Govaerts AS, Buhrer E, Neidhardt EM, Durando X, Baroudjian B, Saiag P, Gaudy-Marqueste C, Ascierto PA, Arance A, Russillo M, Perrot JL, Mortier L, Aubin F, Dalle S, Grange F, Munoz-Couselo E, Mary-Prey S, Amini-Adle M, Mansard S, Lebbe C, Funck-Brentano E, Monestier S, Eggermont AMM, Oppong F, Wijnen L, Schilling B, MandalA M, Lorigan P, van Akkooi ACJ. Combination of encorafenib and binimetinib followed by ipilimumab and nivolumab versus ipilimumab and nivolumab in patients with advanced melanoma with BRAFV600E or BRAFV600K mutations (EBIN): an international, open-label, randomised, controlled, phase 2 study. Lancet Oncol. 2025 Jun;26(6):781-794. doi: 10.1016/S1470-2045(25)00133-0. PMID 40449497